CLINICAL TRIAL: NCT03393741
Title: Pharmacodynamic Biomarkers of Standard Anti-microtubule Drugs as Assessed by Early Tumor Biopsy
Status: Terminated | Type: Observational
Why Stopped: slow accrual
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: UW16151; P30CA014520 (NIH); NCI-2017-01614 (Registry Identifier: NCI Trial ID); 2017-0668 (Other: Institutional Review Board); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison); 1R01CA234904-01 (NIH); Protocol version: 1, 1/6/2017 (Other: UW Madison)
Record Dates: First submitted 2017-11-22; First posted 2018-01-08 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer; Breast Neoplasms
Keywords: Metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — taxane; Paclitaxel; 130-nm albumin-bound paclitaxel; Docetaxel; Vinorelbine; Vinca Alkaloids; ixabepilone; Epothilones; eribulin; Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue samples, pre- and post- 20 hr (+/- 2 hrs) chemotherapy Blood samples, pre- and post- 20 hr (+/- 2 hrs) chemotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Taxane (nab-paclitaxel or paclitaxel): Up to 10 participants will be enrolled on the Taxane arm. The dose and schedule of administration is determined by the treating physician. The first dose will be coordinated in conjunction with research staff who will schedule a research biopsy to be completed on Day 2 of the first planned chemotherapy treatment cycle (C1D2). Participants are not eligible for replacement as long as they are able to have the C1D2 biopsy completed.
  Two tubes of blood of up to 15ml each drawn prior to chemotherapy and again just before or after research biopsy on C1D2. A 15ml sample of blood drawn at the time subject comes off study or at the time of disease progression.
  Tumor core biopsy is obtained as close as possible to 20 hours following initiation of the first planned treatment infusions. Between 2 and 4 cores will be obtained for research biopsy.
  Interventions: Drug: Taxane; Drug: Chemotherapy
- Eribulin: Up to 5 participants will be enrolled on the Eribulin arm. The dose and schedule of administration is determined by the treating physician. The first dose will be coordinated in conjunction with research staff who will schedule a research biopsy to be completed on Day 2 of the first planned chemotherapy treatment cycle (C1D2). Participants are not eligible for replacement as long as they are able to have the C1D2 biopsy completed.
  Two tubes of blood of up to 15ml each drawn prior to chemotherapy and again just before or after research biopsy on C1D2. A 15ml sample of blood drawn at the time subject comes off study or at the time of disease progression.
  Tumor core biopsy is obtained as close as possible to 20 hours following initiation of the first planned treatment infusions. Between 2 and 4 cores will be obtained for research biopsy.
  Interventions: Drug: Eribulin; Drug: Chemotherapy
- Vinorelbine: Up to 5 participants will be enrolled on the Vinorelbine arm. TThe dose and schedule of administration is determined by the treating physician. The first dose will be coordinated in conjunction with research staff who will schedule a research biopsy to be completed on Day 2 of the first planned chemotherapy treatment cycle (C1D2). Participants are not eligible for replacement as long as they are able to have the C1D2 biopsy completed.
  Two tubes of blood of up to 15ml each drawn prior to chemotherapy and again just before or after research biopsy on C1D2. A 15ml sample of blood drawn at the time subject comes off study or at the time of disease progression.
  Tumor core biopsy is obtained as close as possible to 20 hours following initiation of the first planned treatment infusions. Between 2 and 4 cores will be obtained for research biopsy.
  Interventions: Drug: Vinorelbine; Drug: Chemotherapy
- Ixabepilone: Up to 5 participants will be enrolled on the Ixabepilone arm. The dose and schedule of administration is determined by the treating physician. The first dose will be coordinated in conjunction with research staff who will schedule a research biopsy to be completed on Day 2 of the first planned chemotherapy treatment cycle (C1D2). Participants are not eligible for replacement as long as they are able to have the C1D2 biopsy completed.
  Two tubes of blood of up to 15ml each drawn prior to chemotherapy and again just before or after research biopsy on C1D2. A 15ml sample of blood drawn at the time subject comes off study or at the time of disease progression.
  Tumor core biopsy is obtained as close as possible to 20 hours following initiation of the first planned treatment infusions. Between 2 and 4 cores will be obtained for research biopsy.
  Interventions: Drug: Ixabepilone; Drug: Chemotherapy
- Control Arm: Up to 10 participants will be enrolled on the control arm. The dose and schedule of administration is determined by the treating physician. The first dose will be coordinated in conjunction with research staff who will schedule a research biopsy to be completed on Day 2 of the first planned chemotherapy treatment cycle (C1D2). Participants are not eligible for replacement as long as they are able to have the C1D2 biopsy completed.
  Two tubes of blood of up to 15ml each drawn prior to chemotherapy and again just before or after research biopsy on C1D2. A 15ml sample of blood drawn at the time subject comes off study or at the time of disease progression.
  Tumor core biopsy is obtained as close as possible to 20 hours following initiation of the first planned treatment infusions. Between 2 and 4 cores will be obtained for research biopsy.
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Taxane — Taxane is a chemotherapeutic agent and a standard drug for treatment in breast cancer targeting microtubules. This drug is typically infused as a single agent for breast cancer therapy.
  Other Names: paclitaxel; nab-paclitaxel; docetaxel
  Groups: Taxane (nab-paclitaxel or paclitaxel)
Drug: Vinorelbine — Vinorelbine is a chemotherapeutic agent and a standard drug for treatment in breast cancer targeting microtubules. This drug is typically infused as a single agent for breast cancer therapy.
  Other Names: vinca alkaloid
  Groups: Vinorelbine
Drug: Ixabepilone — Ixabepilone is a chemotherapeutic agent and a standard drug for treatment in breast cancer targeting microtubules. This drug is typically infused as a single agent for breast cancer therapy.
  Other Names: epothilone
  Groups: Ixabepilone
Drug: Eribulin — Eribulin is a chemotherapeutic agent and a standard drug for treatment in breast cancer targeting microtubules. This drug is typically infused as a single agent for breast cancer therapy.
  Other Names: halichondrins
  Groups: Eribulin
Drug: Chemotherapy — Chemotherapy is used to treat various stages of breast cancer.

SUMMARY:
Eligible subjects will be assigned to study treatment arms by their treating oncologist, rather than by the study. The drug, dose, and schedule of administration will be determined by the treating physician per NCCN guidelines for standard of care chemotherapy regimens for recurrent or metastatic breast cancer. Study treatment arms include: Taxane (nab-paclitaxel or paclitaxel), Eribulin, Vinorelbine, Ixabepilone, or the control arm (non-microtubule targeted chemotherapies such as doxorubicin, carboplatin, or gemcitabine).

DETAILED DESCRIPTION:
During the screening visit, the following will be taken: medical history; physical exam; ECOG performance status; a pregnancy test if indicated per physician (confirmation of the clinical testing result or assessment of the treating physician whether or not the subject is capable of pregnancy); AST, ALT, CBC (per oncologist); 15 mL blood sample for drug level assessment; 15 mL blood sample for circulating tumor DNA (ctDNA); follow up assessments of cancer; RECIST 1.1 response measurements; and an archived FFPE sample (8 slides) will be obtained.

While enrolled on study, subjects will have the following procedures:

* 15 mL blood sample for drug level assessment on C1D2
* 15 mL blood sample for circulating tumor DNA (ctDNA) on C1D2 and at progression or end of study for a total of 30 mL
* Adverse events related to study procedures (research biopsy & blood draws) will be assessed on C1D2 and at progression or end of study
* Toxicity evaluations will occur throughout the study per the treating MD
* Follow-up assessments of cancer will occur throughout the study per the treating MD
* RECIST 1.1 response measurements will be taken at standard of care imaging
* Fresh biopsy or tumor sampling (4 cores) for analysis of intratumoral drug levels and biomarkers including: markers of proliferation (mitotic index), aneuploidy, and sequencing analysis (ctDNA) on C1D2.

The tests being performed on the samples as part of this study are not investigational.

Subjects will be followed with imaging scans and tumor markers as deemed appropriate by the treating physician. Follow-up scans will be recommended every ~3 cycles as per standard of care. Subjects will be followed for the duration of treatment initiated while taking part in this study. Follow-up will discontinue either 2 months following completion of planned breast cancer treatment or upon the systemic imaging following therapy completion (whichever is later).

ELIGIBILITY:
Inclusion Criteria:

* Men and women with histologically or cytologically demonstrated breast cancer that is deemed metastatic or incurable by the treating physician.
* It is medically appropriate to treat the patient with an antimitotic agent or an intravenous control chemotherapeutic agent by IV infusion at standard doses as per the treating physician. Please see NCCN guidelines for standard of care, p58 for standard chemotherapy regimens for recurrent or metastatic breast cancer7.
* The patient has measureable disease as determined by RECIST 1.1.
* Archived tissue is available from either primary, metastatic site or both.
* It is safe and feasible to obtain a research tumor biopsy on cycle 1 day 2 with a biopsy of an accessible lesion such as liver, lung, lymph node, skin, breast, or bone.
* All pre-chemotherapy test results (tests per treating oncologist discretion) have been reviewed and deemed appropriate for planned chemotherapy by the patient's treating oncologist.

Exclusion Criteria:

* HER2+ breast cancer by standard criteria.
* Pregnant women are excluded from this study because systemic chemotherapy may cause deleterious effects to the fetus. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with systemic chemotherapy, breastfeeding should be discontinued if the mother is enrolled in the trial.
* Planned treatment with hormonal therapy, or targeted oral therapy during trial enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women with metastatic or incurable breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2024-02-11 (Actual); Study Completion 2024-02-11 (Actual)

PRIMARY OUTCOMES:
Feasibility of measuring biomarkers in advanced breast tumors at 20 +/- 2 hours after chemotherapy | Up to 22 hours
  Advanced breast tumors safely sampled and analyzed from 35 subjects.
  In order to successfully test the hypothesis that chromosomal instability in part governs the effect of antimitotic therapies, advanced breast tumors samples must be collected, preserved, and analyzed at 20+/- 2 hours after chemotherapy in order to characterize the effect of the drug on the tumor. A primary question becomes is this process safe and feasible within these time constraints in our clinical setting.

SECONDARY OUTCOMES:
Measure intratumoral drug levels at 20 +/- 2 hours after chemotherapy | Up to 22 hours
  Tumor tissue and plasma samples taken at 20 hours will be assessed for drug levels by the University of Wisconsin 3P Lab.
Measure serum drug levels at 20 +/- 2 hours after chemotherapy | Up to 22 hours
  Tumor tissue and plasma samples taken at 20 hours will be assessed for drug levels by the University of Wisconsin 3P Lab.
Measure PBMC pharmacodynamics at 20 +/- 2 hours after chemotherapy | Up to 22 hours
  Tumor tissue and plasma samples taken at 20 hours will be assessed for drug levels by the University of Wisconsin 3P Lab.
Assess effects of mitosis and DNA damage response at 20 +/- 2 hours after chemotherapy | Up to 22 hours
  Mitotic index will be analyzed by fluorescence in situ hybridization, immunofluorescence, immunohistochemistry, and liquid chromatography and ctDNA
Correlate drug levels and cellular effects with response by RECIST 1:1 to chemotherapy | Up to 2 months following completion of study treatment OR upon the systemic imaging following therapy completion (whichever is later)
  Summary statistics will be used to describe drug levels and cellular effects by response to chemotherapy
Assess genomic profile of metastatic breast cancer | Up to 2 months following completion of study treatment OR upon the systemic imaging following therapy completion (whichever is later)
  This sequencing is measured to understand how changes in treatment response correlate to genomic profile.
Feasibility of quantifying circulating tumor DNA (ctDNA) 20 +/- 2 hours after administration of chemotherapy. | Up to 2 months following completion of study treatment OR upon the systemic imaging following therapy completion (whichever is later)
  This measurement is taken to understand if changes in ctDNA over the stated interval can be correlated to the treatment response and genomic profile from the 35 subjects.
Explore differences in progression free survival (PFS) between chemotherapy arms. | Up to 2 months following completion of study treatment OR upon the systemic imaging following therapy completion (whichever is later)
  PFS will be analyzed using the Kaplan-Meier method and measured from C1D1 until documented progression on imaging scan or death. Patients who do not experience documented progression during the study and are alive at last follow-up will be censored on the date of last imaging scan. Small sample statistical methods will be used to compare PFS curves by chemotherapy arm.
Explore differences in response rate (RR) between chemotherapy arms. | Up to 2 months following completion of study treatment OR upon the systemic imaging following therapy completion (whichever is later)
  Response rate (RR) will be summarized by chemotherapy arm including 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Burkard, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou AS, Tucker JB, Scribano CM, Lynch AR, Carlsen CL, Pop-Vicas ST, Pattaswamy SM, Burkard ME, Weaver BA. Diverse microtubule-targeted anticancer agents kill cells by inducing chromosome missegregation on multipolar spindles. PLoS Biol. 2023 Oct 26;21(10):e3002339. doi: 10.1371/journal.pbio.3002339. eCollection 2023 Oct. PMID 37883329
- See also: UW Carbone Cancer Center home page — http://www.uwhealth.org/cancer